CLINICAL TRIAL: NCT07292194
Title: Pain Experience in Pediatric Patients During Local Anesthesia Infiltration: A Split-Mouth Clinical Trial Comparing Super Pen And Traditional Syringe
Brief Title: Clinical Trial Comparing Pain Perception in Children Using Two Different Local Anesthesia Tools
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lamis D. Rajab (Other)
Responsible Party: Sponsor-Investigator, Lamis D. Rajab, professor, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UJordanLamis2
Record Dates: First submitted 2025-11-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Injection Pain; Local Anesthesia Infiltration; Pediatric Patient
Keywords: clinical trial; split mouth; dental pain; local anesthesia device; local anesthesia infiltration
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super Pen (Active Comparator): Super Pen Computer-controlled Local Anesthesia delivery system
  Interventions: Device: super pen
- Conventional Syringe (No Intervention): Conventional metal syringe

INTERVENTIONS:
Device: super pen — computer controlled local anesthesia delivery device
  Arms: Super Pen

SUMMARY:
The goal of this clinical study is to learn whether the Super Pen (SP) device can reduce pain during local anesthesia (LA) infiltration for primary teeth compared to the conventional syringe (CS) in children aged 6-12 years. It will also explore factors that influence children's pain perception and their preferences for the anesthesia delivery method.

The main questions this study aims to answer are:

* Does the Super Pen (SP) reduce the pain experienced during LA infiltration compared to the conventional syringe (CS)?
* How do factors such as age, sex, and arch treated (maxilla or mandible) influence children's pain perception when using the SP?
* Which method-SP or CS-do children prefer during LA infiltration?

Participants will:

Receive local anesthesia using both the SP and CS techniques in a split-mouth design.

Have their pain responses assessed using self-reported, behavioral, and physiological measures.

Indicate their preference for either technique after both experiences.

DETAILED DESCRIPTION:
This clinical study aims to evaluate and compare the pain perception of pediatric patients aged 6-12 years during local anesthetic (LA) infiltration for primary teeth using the Computer-Controlled Local Anesthetic Delivery (CCLAD) system-Super Pen (SP)-versus the Conventional Syringe (CS) technique. The study follows a split-mouth crossover design, in which each child receives anesthesia using both techniques in separate appointments, allowing for direct within-subject comparison.

Pain assessment will be conducted using a combination of self-reported, behavioral, and physiological measures: the Faces Pain Scale-Revised (FPS-R), the revised Face, Legs, Activity, Cry, Consolability (r-FLACC) behavioral pain scale, and heart rate monitoring. These multiple pain measures used provide a comprehensive evaluation of the child's pain experience.

The study will also investigate the influence of age, sex, and anatomical site (maxilla or mandible) on pain perception during SP administration. In addition, children's preferences for the two delivery systems (SP versus CS) will be recorded after both experiences to assess acceptance and comfort.

The findings of this research aim to contribute to improving pain management strategies in pediatric dentistry, supporting the use of more comfortable and child-friendly anesthesia delivery systems to enhance the dental experience and reduce anxiety in young patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children who were 6-12 years of age, of both sexes.
2. Children who were healthy and medically fit; ASA I .
3. Children who had positive (Class 3) or definitely positive (Class 4) behavior during preoperative behavioral assessments according to the Frankl Scale at the enrollment visit.
4. Children who require bilateral LA infiltration injections for primary teeth, either in the maxilla or mandible, for dental treatment (different types of restoration, stainless steel crowns, pulp therapy, and extractions).
5. Children with positive consent forms approved by their parents/ legal guardians.

Exclusion Criteria:

1. Children who have had a history of unpleasant experiences in medical settings and/or LA injection procedures.
2. Children with any mental, visual, or auditory impairment.
3. Children who have medical or developmentally compromising conditions.
4. Children who had developmental delay problems.
5. Children with a history of chronic disease or use of medication that contraindicate the use of local anesthetics.
6. Children who had active pathosis at the injection site that could affect anesthetic assessment.
7. Patients who have negative (Class 2) or definitely negative (Class 1) behavior during preoperative behavioral assessments according to the Frankl Scale . - -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain using faces pain scale-revised (FPS-r) | Immediately post-procedural (within 1 minute after completion of the local anesthetic injection)
  Pain intensity measured using the Faces Pain Scale - Revised (FPS-R), ranging from 0 to 10, where higher scores indicate greater pain.
Observer-reported pain using Revised Face, Legs, Activity, Cry, Consolability Scale | Periprocedural (during local anesthetic injection, from needle insertion until completion of anesthetic delivery)
  Pain behavior measured using the Face, Legs, Activity, Cry, Consolability - Revised (FLACC-R) Scale, scored from 0 to 10, where higher scores indicate greater pain-related distress.
Physiological-Heart Rate | Baseline (5 minutes prior to local anesthetic injection) and periprocedural (during local anesthetic injection, from needle insertion until completion of anesthetic delivery)
  Changes in heart rate measured in beats per minute (bpm); increases in heart rate indicate higher physiological arousal associated with pain

IPD SHARING:
Plan to Share IPD: Yes